CLINICAL TRIAL: NCT06352216
Title: Prevalence of Synovitis in Adult Patients With Haemophilia A in Germany and Austria
Brief Title: Prevalence of Synovitis in Patients With Haemophilia A
Acronym: SynoPrev
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Principal Investigator, PD Dr. Andreas Strauß, Principal Investigator, University Hospital, Bonn
Other Study IDs: Elo-Ger-2023-1642
Record Dates: First submitted 2024-03-07; First posted 2024-04-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Haemophilia A; Synovitis; Hemophilia Arthropathy; Sonography
Keywords: Synovitis; Haemophilia A; Prevalence
MeSH Terms: conditions — Hemophilia A; Synovitis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Haemophilia A: Patients with severe and moderate Haemophilia A (FVIII < 5 %, ≥ 18 years' old)
  Interventions: Diagnostic Test: Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US); Haemophilia joint health score (HJHS)

INTERVENTIONS:
Diagnostic Test: Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US); Haemophilia joint health score (HJHS) — Each subject is examined for the presence of synovitis using the aforementioned diagnostics.

SUMMARY:
The aim of this study is to evaluate the prevalence of synovitis in adult patients with haemophilia A.

DETAILED DESCRIPTION:
The bleeding disorder haemophilia causes recurrent spontaneous bleedings primarily into the joints and soft tissues. The reason is a congenital lack of factor VIII (haemophilia A) or factor IX (haemophilia B). In Germany, the most affected joints are the ankle, knee, and elbow. The joint bleedings are accompanied by pain and an inflammatory process that leads to synovitis and ultimately to degenerative joint changes resulting in haemophilic arthropathy: The synovial tissue is responsible for removing blood residuals from the joint cavity. However, blood components, especially iron, induce several changes in the synovial tissue. The resulting synovitis leads to damage of cartilage, bone cysts, osteophytes, and joint effusions. Synovitis can even become a bleeding-independent process, especially after repeated bleeding. According to current knowledge, there is no option to prevent synovitis except for preventing bleedings.

In the aftermath of recurrent joint bleedings, various changes in the synovial tissue, the articular cartilage, and the subchondral bone and blood vessels are observed. These changes are accompanied by restricted joint mobility and musculoskeletal dysfunction. In addition to these peripheral structural changes, various studies show that the entire musculoskeletal system is also affected by recurrent joint bleedings, as it adapts to pain.

Improved therapy over the past decades has led to a reduction in major joint bleeding rates. For this reason, it is important to examine whether this has improved the average joint status and how often patients with haemophilia (PwH) are affected by synovitis at all. Sonography is the radiation-free method of choice for the initial determination of synovitis.

In addition to the structural consequences, joint bleedings also lead to pain and reduction in physical performance. When considering the overall process of degenerative joint changes of PwH, it becomes apparent that this also reduces daily mobility and muscle strength. To the best of our knowledge, the effects of the degree of synovitis on pain perception and physical performance have not been evaluated in previous studies.

For this reason, the prevalence of synovitis in PwH and the consequences in relation to the pain situation and physical performance will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participants (≥ 18 years old) suffering from moderate or severe haemophilia A, also with inhibitor or joint replacement
* Complete documentation of hemophilia severity, treatment history (past 12 months), and bleeding events (past 12 months), inhibitor status (at time of enrollment and in past medical history)
* Submitted written consent to participate in the study

Exclusion Criteria:

* Patients suffering from other bleeding disorders conflicting with the research question
* Patients in clinical studies with investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) suffering from moderate (FVIII 1-5 %) or severe (FVIII <1 %) haemophilia A.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Haemophilia early arthropathy detection with ultrasound (HEAD-US) | 20 minutes
  HEAD-US protocol examines both elbow, knee and ankle joints sonographically and assesses the presence of synovitis or joint damage from 0-8 points per joint according to Martinoli et al. 2013. A "total score" of 0 to 48 points is achievable. A higher score means a worse joint status.

SECONDARY OUTCOMES:
The Hemophilia Joint Health Score version 2.1 (HJHS) | 45 minutes
  Clinical joint examination according to De la Corte-Rodriguez et al. 2020. HJHS protocol examines both elbow, knee and ankle joints using a goniometer for range of motion and axial alignment (0-3 points), pain numerical rating scale (0-10 points), swelling (0-3 points), crepitation (0-2 points) and gait abnormalities (0-4 points). A "total score" of 0 to 124 points is achievable. A higher score means a worse joint status.
PROMIS-29 Questionaire | 10 minutes
  Patient-reported outcomes are surveyed using short questionnaires with a stable number of items from seven PROMIS sub scales ("depression", "anxiety", "physical functioning", "impairment due to pain", "fatigue", "sleep impairment", "participation in social roles" and "activities"). The measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  For the sub scales "participation in social roles and activities" and "physical functioning", a high score is interpreted as a good result and for the sub scales "anxiety", "depression", "fatigue", "impairment due to pain", and "sleep impairment" a low score is a good result.
Haemophilia Activities List (HAL) | 10 minutes
  to evaluate to subjective physical performance. A higher scores represent a better functional status.
  Scores can be calculated for each of ten domains of the HAL and a sum score ("Lying / sitting / kneeling / standing" (8-48 Points), "Functions of the legs" (9-54 Points), "Functions of the arms" (4-24 Points), "Use of transportation" (3-18 Points), "Self care" (5-30 Points), "Household tasks" (6-36 Points), "Leisure activities and sports" (7-42 Points), "Upper Extremity Activities" (9-54 Points), "Basic Lower Extremity Activities" (6-36 Points), "Complex Lower Extremity Activities" (9-54 Points), and "Sum score" (42-252 Points).

OTHER OUTCOMES:
Baseline Characteristics | 15 minutes
  1. General anamnesis questionnaire (diseases, pain medication, surgeries, haemophilia related clinical data, date of birth, weight in kilograms, hight in centimeters.
  2. Haemophilia treatment past twelve months (on demand/prophylaxis/non-factor therapy/EHL or SHL therapy)
  3. Bleeding events past twelve months (traumatic or spontaneous)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas C Strauss, PD Dr. med., Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The publication of anonymous patient data is not allowed by informed consent.